CLINICAL TRIAL: NCT03473379
Title: Development and Validation of a Tool for Patient-reported Assessment of Cancer-related Financial Toxicity - Italy
Brief Title: Development and Validation of a Tool for Patient-reported Assessment of Cancer-related Financial Toxicity in Italy
Acronym: PROFTC-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: PROFTC-I
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: economic difficulty, financial toxicity
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase 1: concept elicitation and coding: The aim of this phase is to elicit concepts from patients, caregivers, and oncology clinicians through focus groups of patients and caregivers, qualitative interviews and surveys. Approximately 55 patients or caregivers will participate in this phase.
- Phase 2: Item generation and analysis: The aim of this phase is produce a draft version of the questionnaire. Approximately 90 patients or caregivers will be recruited in this phase for item ranking and analysis through questionnaire evaluation and cognitive interviews.
- Phase 3: Instrument refinement and internal validation: The aim of this phase is generate the final version of the instrument. Approximately 101 patients or caregivers will participate in this phase by completing the questionnaire
- Phase 4: External validation: In this phase the questionnaire will undergo further psychometric testing for validation and approximately 220 patients or caregivers will be asked to complete the PROFTC-I questionnaire along with quality of life instruments

SUMMARY:
The aim of this study is to develop and validate a patient-reported-outcome instrument (PROFTC-I: Patient Reported Outcome Financial Toxicity in Cancer - Italy) able to describe and measure financial problems of Italian patients receiving cancer treatment.

DETAILED DESCRIPTION:
The project will be conducted according to the methodology delineated by the International Society for Pharmacoeconomics and Outcome Research (ISPOR) Patient Reported Outcomes Content Validity Good Research Practices Task Force in the following phases: concept elicitation and coding, item generation and analysis, instrument refinement and internal validation, and external validation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Histologically or cytologically confirmed diagnosis of any type of solid cancer or haematological malignancy
* Written Informed Consent provided
* Medical treatment (chemotherapy, target agents, immunotherapy, hormonal treatment, radiotherapy or combinations of such therapies) ongoing or terminated within the previous 3 months.
* Caregivers of patients who meet the above criteria

Exclusion Criteria:

* Patients with major cognitive dysfunction or psychiatric disorders
* Patients who have never received anticancer medical or radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any type of solid cancer or haematological malignancy who has undergone medical treatment, including chemotherapy, target agents, immunotherapy, hormonal treatment, radiotherapy and combinations of such therapies, or their caregivers, will be recruited in northern, central and southern Italian hospitals..
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Validation of Patient reported outcome financial toxicity of cancer Italian(PROFTC-I) questionnaire | 48 months
  During the development of the questionnaire, individual items (questions), response options, and type of scoring will be determined according to Phases 1-3. Subsequently a principal components analysis (explorative factor analysis) will be done with eigen value set at 1; internal reliability will be assessed by inter-item correlations and Cronbach's alpha ( minimum acceptable 0.70); intraclass correlation coefficient (minimum acceptable 0.80). Correlation of final instrument with the EORTC quality of life questionnaire (criterion validity) will be assessed with using Pearson correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perrone, Principal Investigator — Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale; Jane Bryce, Principal Investigator — Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale; Ciro Gallo, Principal Investigator — University of Campania Luigi Vanvitelli; Silvia Riva, Principal Investigator — St. Mary University, Twickenham, London, GB; Fabio Efficace, Principal Investigator — Northwestern University, Feinberg School of Medicine, GIMEMA,EORTC Quality of Life Group - Rappresentante GIMEMA; Francesco De Lorenzo, Principal Investigator — AIMAC and European Cancer Patient Coalition; Elisabetta Iannelli, Principal Investigator — Segretario Generale FAVO; Laura Del Campo, Principal Investigator — FAVO; Francesca Traclò, Principal Investigator — AIMAC; Massimo Di Maio, Principal Investigator — AO Ordine Mauriziano; Luciano Frontini, Principal Investigator — Federation of Italian Cooperative Oncology Groups; Vincenzo Montesarchio, Principal Investigator — Oncologia, Azienda dei Colli, Napoli - CIPOMO; Lara Gitto, Principal Investigator — Centro per gli Studi Economici e Internazionali - Economic Evaluation & Health Technology Assessment (CEIS EEHTA), Università di Roma "Tor Vergata"; Claudio Jommi, Principal Investigator — Dipartimento di Scienze del Farmaco, Università del Piemonte Orientale; Osservatorio Farmaci, Cergas, SDA Bocconi; Concetta Maria Vaccaro, Principal Investigator — Welfare e Salute CENSIS (Centro Studi Investimenti Sociali), Roma
Locations (5):
- Italy (5):
  - Azienda dei Colli, Napoli
  - Istituto Nazionale Tumori, IRCCS Fondazione Pascale, Napoli
  - Istituto Nazionale Tumori Regina Elena - IRCCS - IFO, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - AO Ordine Mauriziano, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riva S, Arenare L, Di Maio M, Efficace F, Montesarchio V, Frontini L, Giannarelli D, Bryce J, Del Campo L, De Lorenzo F, Iannelli E, Traclo F, Gitto L, Jommi C, Vaccaro CM, Barberio D, Cinieri S, Porta C, Del Mastro L, Zagonel V, Cogoni AA, Bordonaro R, Gimigliano A, Piccirillo MC, Guizzaro L, Gallo C, Perrone F. Cross-sectional study to develop and describe psychometric characteristics of a patient-reported instrument (PROFFIT) for measuring financial toxicity of cancer within a public healthcare system. BMJ Open. 2021 Oct 20;11(10):e049128. doi: 10.1136/bmjopen-2021-049128. PMID 34670762
- [Derived] Riva S, Efficace F, Di Maio M, Bryce J, Del Campo L, De Lorenzo F, Frontini L, Giannarelli D, Gitto L, Iannelli E, Jommi C, Montesarchio V, Traclo F, Vaccaro CM, Arenare L, Canzanella G, Gimigliano A, Romano F, Savio A, Sparavigna L, Piccirillo MC, Guizzaro L, Gallo C, Perrone F. A qualitative analysis and development of a conceptual model assessing financial toxicity in cancer patients accessing the universal healthcare system. Support Care Cancer. 2021 Jun;29(6):3219-3233. doi: 10.1007/s00520-020-05840-z. Epub 2020 Oct 22. PMID 33094357
- [Derived] Riva S, Bryce J, De Lorenzo F, Del Campo L, Di Maio M, Efficace F, Frontini L, Giannarelli D, Gitto L, Iannelli E, Jommi C, Montesarchio V, Traclo F, Vaccaro CM, Gallo C, Perrone F. Development and validation of a patient-reported outcome tool to assess cancer-related financial toxicity in Italy: a protocol. BMJ Open. 2019 Sep 9;9(9):e031485. doi: 10.1136/bmjopen-2019-031485. PMID 31501130